CLINICAL TRIAL: NCT01397019
Title: Chemotherapy for Patients With Locally Advanced Pancreatic Cancer With Additional Chemo-radiotherapy for Patients With Borderline Resectable Tumours
Brief Title: Chemotherapy for Patients With Locally Advanced Pancreatic Cancer (LAPC) With Additional Chemo-radiotherapy (CRT) for Patients With Borderline Resectable Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Per Pfeiffer (Other)
Responsible Party: Sponsor-Investigator, Per Pfeiffer, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPSG 2010-01
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Chemotherapy; Chemoradiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRINOX (Experimental)
  Interventions: Drug: Oxaliplatin, irinotecan, 5-FU & leucovorin

INTERVENTIONS:
Drug: Oxaliplatin, irinotecan, 5-FU & leucovorin — FOLFIRINOX followed by 50 gy/27 F in combination with capecitabine in patients with borderline resectable tumors

SUMMARY:
Treating patients with initial local non-resectable pancreatic cancer with a combination of oxaliplatin, irinotecan & 5-FU(FOLFIRINOX), consolidated with chemoradiotherapy in potentially resectable patients, will result in a high rate of tumor shrinkage allowing subsequent resection in patients with initial borderline resectable tumors and improved overall survival for all patients.

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is the third most common gastrointestinal malignancy and one of the top ten leading causes of cancer deaths in the Western world. Patients with PC can be divided into three subgroups; resectable (rPC), locally advanced (LAPC) and metastatic (mPC). For patients with rPC surgery offers the best chance for long term survival. However it is estimated that only 20% of patients have rPC at the time of diagnosis. For patients with LACP, invasion of local large vessels is most often the cause for non-resectability. The median survival of these patients is between 6 to 12 months and long term survival in is extremely rare. The optimal treatment of LAPC is controversial. Treatment strategies vary between attempts to "downstage" the tumour to rPC, or treat the patients in a palliative setting only. Phase II studies and retrospective series have evaluated various treatments regimens and strategies including chemotherapy and radiotherapy (RT) alone or in combination - chemoradiotherapy (CRT). Results from these trials give no clear answer regarding the best treatment strategy. However, data from several studies shows that treatment of LAPC may result in shrinkage of the tumour, and thus potentially lead to a resection; also data suggests that CRT after chemotherapy improves treatment efficacy. Recent data from patients with mPC has show a combination of oxaliplatin, irinotecan and 5-FU (FOLFIRINOX) increases response rates from 10% to 30% and median survival to 11.1 months. The promising efficacy makes it natural to attempt this treatment in patients with LAPC.

ELIGIBILITY:
Inclusion Criteria: (major)

* non-metastatic pancreatic cancer
* Performance status 0-1
* Bilirubin < 1.5 UNL
* Written informed consent

Exclusion Criteria: (major)

* no prior abdominal radiotherapy
* no prior chemotherapy for pancratic cancer
* no severe comorbidity
* patients must be able to undergo potential abdominal surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
2 year survival rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, Professor, Principal Investigator — Odense University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Herlev University Hospital, Herlev
  - Odense University Hospital, Odense